CLINICAL TRIAL: NCT06154161
Title: Examining the Impact of High-protein Oral Supplement on Protein Status of Adults on Peritoneal Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WheyproteinPD
Record Dates: First submitted 2023-11-21; First posted 2023-12-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Renal Failure; Protein-Energy Malnutrition
Keywords: peritoneal dialysis
MeSH Terms: conditions — Renal Insufficiency; Protein-Energy Malnutrition

STUDY DESIGN:
Intervention Model Description: 6-month prospective interventional clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whey protein consumption (Experimental): Participants will receive 20g total protein of whey protein isolate in 115 mls of water to consume daily for up to 6 months
  Interventions: Dietary Supplement: Whey protein supplement

INTERVENTIONS:
Dietary Supplement: Whey protein supplement — A monthly supply of 35 g of whey protein isolate will be provided to participants in individual sachet packets with instructions of preparation. Every month, participants will come to the center to provide the standard monthly blood sample. At this time, the PI will have participants complete the quality-of-life instrument, ask if there have been any changes in their dietary habits, and collect weights for up to 6-months. Additionally, participants will indicate if they had consumed the protein daily and/or bring back their empty/full satchel packets. As this is a feasibility trial, it is necessary to determine the compliancy of consuming protein daily and the amount. Furthermore, understanding how protein markers may be affected by consumption of the protein daily vs less frequently throughout the week is important to establish improved recommendations for consumption of protein supplements.

SUMMARY:
This is a 6-month prospective interventional clinical trial designed to evaluate the impact of whey protein isolate oral supplement on protein status. Differences in protein status will be evaluated with review of the medical chart from standard of care monthly blood collection for serum albumin, total protein, and normalized protein catabolic rate (nPCR) as detected by serum urea nitrogen. Mid-arm circumference and weight will be measured to ensure no significant changes. Quality of life will be measured to detect if the addition of protein aided in overall quality of life. There will be a 3-month recruitment period prior to the start of the trial to ensure the potential participants are familiarized with the clinical trial. After the recruitment period has finished, eligible participants will sign the consent form in order to participate in the study. At this point, participants will be provided the supplements for the month and instructed with the amount of water and how to mix with the provided measuring and drinking cup.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* diagnosed with stage 5 Chronic Kidney Disease for at least 3 months prior to the starting date of the trial
* on peritoneal dialysis at least three months prior to the starting date of the trial
* can provide signed informed consent
* have no dietary restriction
* no food allergies
* no chewing/swallowing difficulties.

Exclusion Criteria:

* not meeting the above
* pregnant/lactating as either self-reported or determined by the medical director

  * Chronic Kidney Disease patient stages 1-4.
  * Chronic Kidney Disease patient undergoing hemodialysis.
* use of other protein supplement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Serum albumin | up to 6 months of the study
  Collection of serum albumin to identify a change from pre-post to analyze the effect protein isolate had on inflammation marker and protein status.

SECONDARY OUTCOMES:
Total protein | up to 6 months of the study
  Collection of whole blood total protein to identify a change from pre-post to analyze the effect protein isolates had on protein stores.
normalized protein catabolic rate (nPCR) | up to 6 months of the study
  Collection of nPCR through serum to identify a change from pre-post to analyze the effect protein isolates had on nPCR.
mid-arm muscle circumference | up to 6 months of the study
  measuring mid-arm circumference from baseline to the end of the study to determine that protein isolates did not affect muscle mass.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette M Andrade, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - UF Health Dialysis Center, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No
Data and files will be secured in locked filling cabinets and office space. Paper questionnaires will only include date and research study assigned participant number. Data that is originally captured as hardcopy/paper (e.g. questionnaires) will be transcribed to encrypted electronic files.
  Following the completion of the study, any potential identifiers will be removed from data to meet HIPAA de-identification standards (According to the October 2002 Privacy Rule § 164.514.(b).2. the indicated information/will be removed from all study records).
  Upon publication, de-identified data can be shared with other researchers.